CLINICAL TRIAL: NCT04177771
Title: A Prospective Randomized Controlled Multi-center Clinical Study to Evaluate The Safety and Effectiveness of The RxSight Light Adjustable Lens (LAL) In Subjects Desiring an Extended Depth of Focus
Brief Title: A Clinical Study to Evaluate The Safety and Effectiveness of The RxSight Light Adjustable Lens (LAL) In Subjects Desiring an Extended Depth of Focus
Status: Terminated | Type: Interventional
Why Stopped: Technology changes.
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-033
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Aphakia; Cataract; Presbyopia
Keywords: Light Adjustable Lens; Intraocular lens; LAL
MeSH Terms: conditions — Aphakia; Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to undergo experimental or control treatment.
Who Masked: Outcomes Assessor
Masking Description: Select post operative assessments will be performed on both the experimental and control treatment groups by an examiner who will be masked to the treatment group assignments.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Light adjustable lens (LAL) and Light Delivery Device (LDD) (Experimental)
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population
- SofPort LI61AO IOL (Active Comparator)
  Interventions: Device: SofPort LI61AO IOL; Device: Tecnis ZCB00 or ZTC150 IOL

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population — Experimental treatment group will receive Light adjustable lens with Light delivery Device treatments
  Arms: Light adjustable lens (LAL) and Light Delivery Device (LDD)
Device: SofPort LI61AO IOL — Control treatment group will receive SofPort LI61AO IOL
  Arms: SofPort LI61AO IOL
Device: Tecnis ZCB00 or ZTC150 IOL — Control treatment group will receive Tecnis ZCB00 or ZTC150 IOL
  Arms: SofPort LI61AO IOL

SUMMARY:
The primary objective of this study is to evaluate, for the visual correction of aphakia and presbyopia, the safety and effectiveness of the RxSight Light Adjustable Lens (LAL) to provide an extended depth of focus (improve intermediate and near visual acuity without compromising distance visual acuity) in subjects who have undergone bilateral implantation with the LAL and subsequent light treatments for refractive and presbyopia correction (LAL group).

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for the bilateral implantation of either the LAL or SofPort LI61AO intraocular lens (IOL) (Bausch + Lomb).
* Must be willing to be randomized to either the LAL group (bilaterally implanted with the LAL and receive light treatments for refractive and presbyopia correction) or the Control group
* Between the ages of 40 and 80 inclusive on the day the cataract surgery is performed.
* Cataractous lens changes as demonstrated by best corrected distance visual acuity (BCDVA) of 20/40 or worse with or without a glare source in both eyes.
* Willing and able to comply with the requirements for study specific procedures and visits.
* Able to complete a written questionnaire in English.

Exclusion Criteria:

* Pre-existing macular disease in either eye.
* Patient with sufficiently dense cataract that precludes examination of the macula in either eye.
* Diabetes with any evidence of retinopathy in either eye.
* Evidence of glaucomatous optic neuropathy in either eye.
* History of uveitis in either eye.
* Keratoconus or suspected of having keratoconus in either eye.
* Has undergone previous corneal or intraocular surgery in either eye, except eyes with previous pterygium excision are permitted as long as the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Subjects taking systemic medication that may increase sensitivity to UV light such as tetracycline, doxycycline, psoralens, amiodarone, phenothiazines, chloroquine, hydrochlorothiazide, hypericin, ketoprofen, piroxicam, lomefloxacin, and methoxsalen. LDD treatment in patients taking such medications may lead to irreversible phototoxic damage to the eye. This is only a partial list of photosensitizing medications. Please evaluate all medications that the patient is taking for this effect prior to consideration for implantation.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* History of ocular herpes simplex virus in either eye.
* Subject who has participated within another ophthalmic clinical trial within the last 3 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vold Vision, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Light Adjustable Lens (LAL) and Light Delivery Device (LDD); Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population: Light Adjustable lens (LAL) and Light Delivery Device (LDD): Experimental treatment group will receive Light adjustable lens with Light delivery Device treatments
- Tecnis ZCB00 or ZTC150 IOL: Tecnis ZCB00/ZTC150 IOL: Control treatment group will receive Tecnis ZCB00 or ZTC150 IOL
Period: Pre-COVID Population
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL
Started | 10 | 7 (1 subject received the ZCB00 IOL in their primary eye and the ZTC150 IOL in their fellow eye. The 6 other subjects all received the ZCB00 IOL bilaterally.) | 0 | 0
Completed | 10 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Modified Safety Population
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL
Started | 0 | 0 | 7 | 10
Completed | 0 | 0 | 7 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to the COVID-19 pandemic, study visits for the first 17 subjects enrolled (Light adjustable lens (LAL) and Light Delivery Device (LDD) - Pre-COVID population and Tecnis ZCB00 or ZTC150 IOL) may have been delayed outside protocol specified windows or missed completely. Per the protocol, these subjects will be excluded from the Full Analysis Set populations.
Groups:
- Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population; Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population: Light Adjustable lens (LAL) and Light Delivery Device (LDD): Experimental treatment group will receive Light adjustable lens with Light delivery Device treatments
- Total: Total of all reporting groups
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL | Total
Number analyzed (Participants) | 10 | 7 | 7 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.7) | 69.2 (5.5) | 65.4 (8.5) | 66.6 (5.5) | 66.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 3 | 7 | 23
  Male | 0 | 4 | 4 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 | 0 | 7
  Not Hispanic or Latino | 6 | 5 | 6 | 10 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 9 | 7 | 7 | 10 | 33
  Race: Black/African American | 1 | 0 | 0 | 0 | 1
  Race: Asian | 0 | 0 | 0 | 0 | 0
  Race: American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0
  Race: Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Other | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular Depth of Focus (DOF) Measured at the logMAR 0.2 Level Compared Between LAL Treatment Group and Control Group
Description: Comparison of monocular distance visual acuity (VA) in logMAR, measured with different spherical lens powers over the eye. The lens diopter value corresponding to the intercepted point of the 0.20 logMAR visual acuity was determined by interpolation for each group mean. The DOF at Postop Month 6 was the absolute difference between the negative lens diopter value corresponding to the 0.20 logMAR visual acuity and 0 diopter for each group.
Time Frame: Postop Month 6
Measure: Number; unit: Diopters
Units Other Than Participants: Primary Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL
Number analyzed (Participants) | 10 | 7 | 7 | 10
Number analyzed (Primary Eyes) | 10 | 7 | 7 | 10
Diopters | 2.30 | 0.97 | 1.58 | 0.85

2. Primary Outcome: Monocular Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) at 67 cm Compared Between LAL Treatment Group and Control Group
Description: Comparison of monocular Distance-Corrected Intermediate Visual Acuity measured at 67 cm between LAL treatment and control groups
Time Frame: Postop Month 6
Population: Since the sample sizes of each group did not meet the minimum requirements (8 eyes per lens group) for statistical power per study protocol, a mean difference comparison test was not performed. 95% confidence intervals were calculated and compared between groups.
Measure: Mean (95% Confidence Interval); unit: LogMAR
Units Other Than Participants: Primary Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL
Number analyzed (Participants) | 10 | 7 | 7 | 10
Number analyzed (Primary Eyes) | 10 | 7 | 7 | 10
LogMAR | 0.09 [-0.02 to 0.19] | 0.29 [0.13 to 0.44] | 0.13 [0.01 to 0.26] | 0.33 [0.21 to 0.46]

3. Primary Outcome: Outcome of Monocular Photopic DCIVA at 67 cm Better Than or Equal to 0.20 logMAR for the LAL Group at Postop Month 6
Description: Percent of LAL treatment group with monocular Distance-Corrected Intermediate Visual Acuity measured at 67 cm better than or equal to 0.20 logMAR
Time Frame: 6 months
Population: Due to the COVID-19 pandemic, study visits for the first 17 subjects enrolled (Light adjustable lens (LAL) and Light Delivery Device (LDD) - Pre-COVID population and TECNIS ZCB00 or ZTC150 IOL) may have been delayed outside protocol specified windows or missed completely. Since the sample sizes of each group did not meet the minimum requirements (28 eyes per lens group) for statistical power per study protocol, 95% confidence intervals were calculated.
Measure: Number (95% Confidence Interval); unit: percentage of Primary Eyes
Units Other Than Participants: Primary Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population
Number analyzed (Participants) | 10 | 7
Number analyzed (Primary Eyes) | 10 | 7
percentage of Primary Eyes | 80 [44.4 to 97.5] | 71.4 [29.0 to 96.3]

4. Primary Outcome: Monocular Photopic Best Corrected Distance Visual Acuity (BCDVA) Compared Between LAL Treatment Group and Control Group
Description: Comparison of monocular Best-Corrected Distance Visual Acuity between LAL treatment and control groups
Time Frame: Postop Month 6
Population: Since the sample sizes of each group did not meet the minimum requirements (42 eyes per lens group) for statistical power per study protocol, a mean difference comparison test was not performed. 95% confidence intervals were calculated and compared between groups.
Measure: Mean (95% Confidence Interval); unit: LogMAR
Units Other Than Participants: Primary Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL
Number analyzed (Participants) | 10 | 7 | 7 | 10
Number analyzed (Primary Eyes) | 10 | 7 | 7 | 10
LogMAR | 0.00 [-0.08 to 0.09] | -0.11 [-0.16 to -0.05] | 0.02 [-0.09 to 0.12] | -0.06 [-0.13 to 0.01]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Due to the COVID-19 pandemic, study visits for the first 17 subjects enrolled may have been delayed outside protocol specified windows or missed completely (i.e., "Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population", "Tecnis ZCB00 or ZTC150 IOL"). Per the protocol, these subjects will be excluded from the Full Analysis Set populations.
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population | Tecnis ZCB00 or ZTC150 IOL | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population | SofPort LI61AO IOL
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/7 | 1/7 | 1/10
Other Adverse Events (participants affected / at risk) | 9/10 | 2/7 | 4/7 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population (N=10) | Tecnis ZCB00 or ZTC150 IOL (N=7) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population (N=7) | SofPort LI61AO IOL (N=10)
Gall bladder removal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laparoscopic cholecystectomy for gall stones (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Internal and external hemorrhoids requiring hospitalization (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Pre-COVID Population (N=10) | Tecnis ZCB00 or ZTC150 IOL (N=7) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) - Modified Safety Population (N=7) | SofPort LI61AO IOL (N=10)
Primary and Fellow Eye, BCDVA letter drop 10 letters or worse compared to week 3 (Eye disorders) | 5 (8) | 1 (1) | 3 (5) | 0 (0)
Primary and Fellow Eye, Posterior capsular opacity requiring YAG (Eye disorders) | 5 (8) | 1 (2) | 3 (5) | 1 (2)
Primary and Fellow Eye, Non-clinically significant cystoid macular edema (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Primary and Fellow Eye, Punctate Epithelial Erosion causing watery and uncomfortable eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary and Fellow Eye, Subjective symptom of blurry vision, red in lights and starbursts (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Primary and Fellow Eye, Subjective symptom of much less crisp vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Primary and Fellow Eye, Glare or halos or double/multiple images (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Primary and Fellow Eye, Drusen (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Primary and Fellow Eye, Cellulitis, hordeolum (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, study visits for the first 17 subjects enrolled may have been delayed outside protocol specified windows or missed completely. Per the protocol, these subjects will be excluded from the Full Analysis Set populations. Based on the sample size calculations, at least 42 subjects per lens group with available monocular photopic BCDVA and DCIVA for the primary eyes at Postop Month 6 were needed; however, the sample size was too small to analyze these endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT04177771/Prot_SAP_001.pdf